CLINICAL TRIAL: NCT04375371
Title: Klinische Und Metabolische Charakterisierung Der Langzeitverläufe Von Adipositas-Patienten Mit Vergleich Von Bariatrisch Operierten zu Nicht Operierten Patienten
Brief Title: Clinical and Metabolic Characterization of Long-term Courses of Obesity Patients
Acronym: AdipFollowup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 338/2019BO1
Record Dates: First submitted 2019-10-18; First posted 2020-05-05 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2020-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese patients who have received a bariatric surgery (Active Comparator): Obese patients who have undergone a bariaric surgery as part of routine clinical management within the indication of this intervention.
  Interventions: Procedure: Bariatric surgery
- Obese patients without a bariatric surgery (No Intervention): Obese patients who have not undergone bariaric surgery.

INTERVENTIONS:
Procedure: Bariatric surgery — Obese patients who haveundergone bariatric surgery as part of routine clinical management within the indication of this intervention.
  Arms: Obese patients who have received a bariatric surgery

SUMMARY:
The long-term courses after bariatric surgery are not sufficiently known. Furthermore there is a heterogeneity in postoperative responses.

The aim of this study is to investigate the glycemic course (prediabetes, development of diabetes) of patients with obesity (BMI>=35 kg/m2) who had undergone bariatric surgery compared to patients with obesity who have not. A further aim is to investigate predictors of weight development, development of body composition and insulin sensitivity of patients who had undergone bariatric surgery compared to obesity patients who have not undergone bariatric surgery. The long-term courses after different surgical procedures (Roux-Y vs Sleeve) will be compared.

In this study 300 patients with obesity who had been metabolically characterized in a previous study will be recruited.

These patients are examined (medical history, physical examination including ECG, BIA, weight, height) and metabolically characterized.

Participants without diabetes undergo a glucose tolerance test and fasting blood sampling will be performed in participants with diabetes. All patients complete questionnaires to activity, nutrition, life quality, impulsiveness, depression and eating behavior.

Randomly selected participants will be offered an abdominal fat tissue biopsy. When consent is given, this will be performed at least two days after the glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the study " Das ADIP-Programm: Charakterisierung adipöser Probanden mittels genauer phänotypischer und genotypischer Klassifizierung"

Exclusion Criteria:

* BMI < 35 kg/m2 at start of the previous study
* Women during pregnancy and lactation
* Patients who are unable to give their consent
* Patients who have undergone surgery within the last 3 months
* acute disease or infection within the last 4 months
* HIV- or hepatitis B/C-positive
* for biopsy of fat tissue: known coagulation disorder or PTT or INR out of reference range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of diabetes | On average 11 years after baseline assessment (previous study).
  Diabetes mellitus as determined by HbA1c, fasting glucose and/or post-challenge glucose (120 min after an 75g oral glucose tolerance test).
Incidence of prediabetes | On average 11 years after baseline assessment (previous study).
  Prediabetes as determined by fasting glucose and/or post-challenge glucose (120 min after an 75g oral glucose tolerance test).

SECONDARY OUTCOMES:
Change in body weight | Baseline (previous study) and after an average of 11 year (follow-up visit)
  Effect of bariatric surgery versus no surgery on body weight assessed by calculating BMI.
Change in body fat mass | Baseline (previous study) and after an average of 11 year (follow-up visit)
  Effect of bariatric surgery versus no surgery on body fat mass assessed by bioelectric impedance analysis.
Change in fat free mass | Baseline (previous study) and after an average of 11 year (follow-up visit)
  Effect of bariatric surgery versus no surgery on fat free (kg) mass assessed by bioelectric impedance analysis.
Change in insulin sensitivity | Baseline (previous study) and after an average of 11 year (follow-up visit)
  Effect of bariatric surgery versus no surgery on insulin sensitivity assessed by 75g oral glucose tolerance test.
Occurence of diabetic complications - nephropathy | On average 11 years after baseline assessment (previous study).
  Occurence of diabetes complications: nephropathy measured as urine microalbuminuria.
Occurence of diabetic complications - retinopathy | On average 11 years after baseline assessment (previous study).
  Occurence of diabetes complications: retinopathy assessed by retinal examination
Occurence of diabetic complications - neuropathy | On average 11 years after baseline assessment (previous study).
  Occurence of diabetes complications: neuropathy assessed by Michigan-neuropathy screening tool
Occurence of macrovascular complications | On average 11 years after baseline assessment (previous study).
  Occurence of manifestations of coronary artery disease (myocardial infarction, angina pectoris) or stroke or peripheral artery disease.

OTHER OUTCOMES:
Occurene of depressions | On average 11 years after baseline assessment (previous study).
  Occurene of depressions as estimate of quality of life assessed by the BDI-II Beck's Depression Inventory (BDI-II) questionnaire (minimum value:0, maximum value: 63; higher score indicate more severe depressive symptoms).
impulsivity measurement | On average 11 years after baseline assessment (previous study).
  Impulsivity assessed by the Barratt Impulsiveness Scale-15 (BIS-15) questionnaire (minimum value:15, maximum value: 60; higher score indicate higher impulsivity).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wagner, PD Dr., Principal Investigator — University of Tuebingen, Department of Internal Medicine IV
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No